CLINICAL TRIAL: NCT00528242
Title: A Randomized, Double Blind, Placebo-controlled, Cross-over Pilot Study to Examine the Safety, Tolerability and Pharmacodynamic Profile of Repeat Oral Doses of SLx-2101 Once Daily for up to 14 Days in Subjects With Secondary Raynaud's Disease.
Brief Title: Safety, Tolerability, and Pharmacodynamic Profile of Oral 2101 in Secondary Raynaud's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Response Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SLx-2101-07-04
Record Dates: First submitted 2007-09-11; First posted 2007-09-12 (Estimated); Last update posted 2023-11-18 (Actual); Status verified 2015-01

CONDITIONS: Raynaud's Disease
MeSH Terms: conditions — Raynaud Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): SLx-2101
  Interventions: Drug: SLx-2101
- 2 (Placebo Comparator): Matching Placebo Dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SLx-2101
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
To investigate the severity of secondary Raynaud's disease-related attacks during the 14 days 2101 dosing period.

DETAILED DESCRIPTION:
1. Number and cumulative duration of Raynaud's attacks.
2. Adverse events and changes in vital signs.
3. SLx-2101 pharmacokinetic parameters derived after dosing on Day 1 and Day maximum plasma concentration (Cmax), area under the plasma concentration-time curve (AUC0-4), time to Cmax (tmax), and accumulation ratio

ELIGIBILITY:
Inclusion Criteria:

* male and female ages 18 and 65 y.o.
* BMI Body weight within a body mass index range of 17 - 30 kg/m2 (inclusive).

Exclusion Criteria:

* Hypersensitivity to the active substance of SLx-2101or to any of the excipients.
* Past or present disease that is judged by the Investigator to have the potential to interfere with the study procedures, compromise safety, or affect the pharmacokinetic and pharmacodynamic evaluations

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2007-06; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Raynaud's condition scores after 14 days of SLx-2101 | 14 days

SECONDARY OUTCOMES:
Safety and tolerability | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: M Baumaker, MD, Study Director — University des Saarlandes
Locations (1):
- University des Saarlandes, Homburg, Germany